CLINICAL TRIAL: NCT04219904
Title: Evaluation of Resectable Cervical Carcinoma With PET/MRI
Brief Title: PET/MRI Scan for the Evaluation of Resectable Stage IA1-IB3 Cervical Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-0066; NCI-2019-08255 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0066 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Stage IA Cervical Cancer; Stage IA1 Cervical Cancer; Stage IA2 Cervical Cancer; Stage IB Cervical Cancer; Stage IB1 Cervical Cancer; Stage IB2 Cervical Cancer; Stage IB3 Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Fluorodeoxyglucose F18; gadobutrol; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (PET/MRI) (Experimental): Patients receive fludeoxyglucose F-18 and gadobutrol IV over 1 minute and undergo PET/MRI over 90-120 minutes.
  Interventions: Other: Fludeoxyglucose F-18; Drug: Gadobutrol; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Gadobutrol — Given IV
  Other Names: BAY86-4875; Gadavist; Gadograf; Gadovist; Protovis; ZK 135079
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well positron emission tomography/magnetic resonance imaging (PET/MRI) scan works in checking patients with stage IA1-IB3 cervical cancer that can be removed by surgery (resectable). PET/MRI scan may help doctors learn more about the spread of the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess depth of cervical invasion with positron emission tomography/magnetic resonance imaging (PET/MRI) in patients with cervical cancer in clinical Federation of Gynecology and Obstetrics (FIGO) staging undergoing evaluation for surgical resection and correlate with pathology.

SECONDARY OBJECTIVES:

I. To correlate lymph node involvement on PET/MRI with pathology. II. To assess the inter-observer variability in the interpretation of PET/MRI. III. To correlate the quantitative imaging parameters of the tumor, such as the volumetric size, blood oxygen level dependent (BOLD), intravoxel incoherent motion (IVIM) analysis, apparent diffusion coefficient (ADC), diffusion tensor imaging (DTI), dynamic contrast-enhanced (DCE), metabolic tumor volume (MTV), total lesion glycolysis (TLG), standardized uptake value (SUV) and the glucose metabolic rate (GMR) with lymphovascular space invasion (LVSI) and tumor grade on surgical pathology.

OUTLINE:

Patients receive fludeoxyglucose F-18 and gadobutrol intravenously (IV) over 1 minute and undergo PET/MRI over 90-120 minutes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with suspected clinical stage IA1-IB3 cervical cancer except patients with tumors > 4 cm
* No contraindications to MRI
* Patients undergoing surgical procedure at MD Anderson
* Suspected cervical cancer

Exclusion Criteria:

* Patients who have contraindication to MRI
* Glomerular filtration rate (GFR) < 30
* Pregnant patients
* Patients with history of previous radiation
* Patients with previous surgery for cervical cancer, unless residual tumor noted on physical exam
* Patients with endometrial cancer extending to the cervix
* Allergic reaction to gadolinium based contrast
* Body weight of greater than 450 (181.4 kg)
* Patients requiring general sedation
* Extremely claustrophobic patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of diagnosing depth of invasion on positron emission tomography/magnetic resonance imaging (PET/MRI) | 3 years
  Both PET/MRI and pathology results will be dichotomized into binary outcomes and the accuracy of PET/MRI will assessed.

SECONDARY OUTCOMES:
Assessing the Lymph node involvement by PET/MRI | 3 years
  Will determine the relationship with pathology.
Inter-observer variability of PET/MR | 3 years
  A PET report for clinical use will be generated by a radiologist with appropriate training and credentialing to read PET images. A separate MRI report for clinical use will be generated by a radiologist with appropriate training and credentialing to read MRI. Subsequently, PET/MR images will be evaluated by two radiologists who have appropriate training to read both PET and MRI and 2 research reports will be generated. Inter-observer variability of PET/MRI will be calculated using Cohen's kappa coefficient.
Quantitative imaging parameters of the tumor | 3 years
  Correlate the quantitative imaging parameters of the tumor, such as the volumetric size, blood oxygen level-dependent (BOLD), apparent diffusion coefficient (ADC), IVIM analysis, diffusion tensor imaging (DTI), dynamic contrast-enhanced (DCE), MTV, TLG, standardized uptake value (SUV) and GMR with LVSI and tumor grade on surgical pathology which serves as gold standard. Two-sample t-test or analysis of variance (ANOVA) will be used for comparing the group means between LVSI positive/negative groups and among tumor grades and types. Other statistical analysis will be carried out as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Sanaz Javadi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org